CLINICAL TRIAL: NCT01536743
Title: A Open Label Phase II Study of the Efficacy and Safety of PD0332991 a Selective Inhibitor of the Cyclin Dependent Kinases 4 and 6 in Patients With Recurrent Ovarian Cancer Demonstrating Rb-proficiency and Low p16 Expression
Brief Title: A Open Label Study of the Efficacy and Safety of PD0332991 a Selective Inhibitor of the Cyclin Dependent Kinases 4 and 6 in Patients With Recurrent Ovarian Cancer Demonstrating Rb-proficiency and Low p16 Expression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-003234
Record Dates: First submitted 2011-12-01; First posted 2012-02-22 (Estimated); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Ovarian Epithelial Carcinoma
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PD0332991 (Experimental): 30 patients with recurrent ovarian epithelial carcinoma demonstrating Rb-proficiency and absent or low expression of p16 will be registered to receive PD0332991 once a day by mouth in the morning on an empty stomach.
  PD0332991 will be administered daily for 3 weeks followed by 1 week off treatment (28 day cycle).
  Interventions: Drug: PD0332991

INTERVENTIONS:
Drug: PD0332991 — 30 patients with recurrent ovarian epithelial carcinoma demonstrating Rb-proficiency and absent or low expression of p16 will be registered to receive PD0332991 once a day by mouth in the morning on an empty stomach.
  PD0332991 will be administered daily for 3 weeks followed by 1 week off treatment (28 day cycle).

SUMMARY:
The purpose of this study is to obtain an estimate of the biochemical response rate as determined by CA125 response using the Gynecologic Cancer Intergroup (GCIG) response criteria of PD0332991 in patients with recurrent ovarian epithelial carcinoma. CA125 response is defined as ≥ 50% decrease from the baseline CA125 level and confirmed ≥ 21 days after initial evaluation (baseline is defined as the higher value of 2 pre-treatment CA125 assessments).

ELIGIBILITY:
Inclusion Criteria

1. Histologically-confirmed ovarian epithelial (including fallopian tube and primary peritoneal) carcinoma.
2. 2. Baseline paraffin embedded tissue from the patient's primary diagnosis is requested before study enrolment and should be forwarded to the designated central laboratory where central assessment of Rb and p16 expression will be performed by using immunohistochemistry. In patients with measurable disease a tissue biopsy may be obtained by core biopsy and submitted to the designated central laboratory.
3. GCIG-defined CA125 progression and absence of disease upon imaging or small-volume asymptomatic disease upon imaging and who have progressed following one, two or three lines of chemotherapy for recurrent disease.
4. If patients have small-volume disease the current study will be restricted to patients with minimal ascites not causing abdominal distention/mesenteric thickening or not requiring paracentesis, or lesions ≤4 cm by spiral computed tomography [CT] or magnetic resonance imaging [MRI] at baseline.
5. Two pretreatment CA125 values (documented on two occasions taken at least one week apart) must be at least twice the upper limit of normal, or twice the nadir value if pretreatment CA125 values never normalized.
6. Patients with platinum-sensitive or platinum-resistant disease defined by recurrence or progression of disease > 6 months or ≤ than 6 months after completion of frontline platinum based chemotherapy.
7. ECOG performance status ≤ 1 and patients are to be ≥21 years of age.
8. Resolution of any toxic effects of prior therapy (except alopecia) to NCI CTCAE v.3.0 Grade ≤ 1 and to baseline laboratory values as defined in the inclusion criterion immediately below.
9. Adequate organ and bone marrow function as evidenced by:

   * hemoglobin ≥ 9.0 g/dL
   * absolute neutrophil count ≥ 1.5 x 109/L
   * platelet count ≥ 100 x 109/L
   * Renal function, as follows:
   * Serum creatinine ≤ 1.5 x the ULN or calculated creatinine clearance ≥ 40 mL/min
   * AST and ALT ≤ 2.5 x ULN
   * total bilirubin ≤ 1.5 x ULN unless increase is due to Gilbert's disease or similar syndrome involving slow conjugation of bilirubin,
10. Adequate coagulation parameters (within 21 days prior to registration), International Normalized Ratio (INR) ≤1.5; Activated ProThrombin Time (APTT) ≤ 1.5 x ULN.
11. Patient must be willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
12. Informed consent must be obtained in writing for all patients prior to performing study/screening procedures and prior to registration into the study.

Exclusion Criteria

Patients presenting with any of the following will not be included in the study:

1. More than 4 prior chemotherapy regimens in the treatment of ovarian cancer.
2. Anticipation of immediate need for a major surgical procedure (e.g., impending bowel obstruction, gastrointestinal perforation) or radiation therapy during the trial.
3. Diagnosis of any second malignancy within the last 5 years, except for adequately treated basal cell or squamous cell skin cancer, or for in situ carcinoma of the cervix uteri or breast.
4. Treatment with chemotherapy, radiotherapy, surgery, blood products, or an investigational agent within 3 weeks of trial enrolment.
5. Any of the following within 6 months prior to trial registration: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, NYHA class III or IV congestive heart failure, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis, or other thromboembolic event. PD0332991 in Recurrent Ovarian Cancer
6. History of brain metastases, spinal cord compression, or carcinomatous meningitis.
7. Patient of child-bearing potential is evidently pregnant (eg, positive human chorionic gonadotropin test) or is breast feeding. A woman with child bearing potential is defined as not surgically sterile or being post-menopausal for less than 6 months.
8. Patient of child-bearing potential is not willing to use adequate contraceptive precautions. Adequate effective method of contraception are those which result in low failure rates, less than 1% per year, such as non-hormonal IUD, condoms, sexual abstinence or vasectomised partner.
9. Known active infection, or on antiretroviral therapy for HIV disease or positive test for chronic hepatitis B or C infection.
10. Mental condition rendering the patient unable to understand the nature, scope, and possible consequences of the trial.
11. Refusal or inability to give informed consent to participate in the trial.
12. Corrected QT (QTc) interval >470 msec.
13. If radiotherapy is required in a given patient, that patient should be withdrawn from the study.
14. Current use or anticipated need for: Food or drugs that are known strong CYP3A4 inhibitors (i.e. grapefruit juice, verapamil, ketoconazole, miconazole, itraconazole, posaconazole, erythromycin, clarithromycin, telithromycin, indinavir, saquinavir, ritonavir, nelfinavir, lopinavir, atazanavir, amprenavir, fosamprenavir, nefazodone, diltiazem, and delavirdine.
15. Other severe acute or chronic medical or psychiatric condition, or significant laboratory abnormality requiring further investigation that may cause undue risk for the patient's safety, inhibit protocol participation, or interfere with interpretation of trial results, and in the judgment of the investigator would make the patient inappropriate for entry into this trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-12-15 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
Estimate biochemical response rate as determined by CA125 response using the Gynecologic Cancer Intergroup (GCIG) response criteria of PD0332991 in patients with recurrent ovarian epithelial carcinoma. | 4 weeks
  CA125 response is defined as ≥ 50% decrease from the baseline CA125 level and confirmed ≥ 21 days after initial evaluation (baseline is defined as the higher value of 2 pre-treatment CA125 assessments).

SECONDARY OUTCOMES:
Toxicity of PD0332991. | 4 weeks
  Toxicity of PD0332991 will be graded using the NCI Common Toxicity Criteria, version 3.0
Assess health-related quality of life (HRQL), | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gottfried Konecny, M.D., Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States